CLINICAL TRIAL: NCT02877147
Title: The Evaluation of the Summer Electronic Benefits for Children Demonstration
Brief Title: The Evaluation of the Summer EBT for Children Demonstration
Acronym: SEBTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abt Associates (Industry)
Collaborators: Maxiumus (Unknown); USDA Food and Nutrition Service (U.S. Federal Agency); Mathematica Policy Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17322
Record Dates: First submitted 2016-08-16; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Food Insecurity Among Children; Dietary Modification
MeSH Terms: interventions — Food Assistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- $60 SEBTC Benefit Group (Experimental): Households received $60 per summer month when school was not in session for each eligible child (Summers 2011-2013).
  Interventions: Other: SEBTC
- $30 SEBTC Benefit Group (Experimental): Households received $30 per summer month when school was not in session for each eligible child (Summer 2013 only).
  Interventions: Other: SEBTC
- No Intervention Group (No Intervention): Households with eligible children were not issued SEBTC benefits (Summers 2011 and 2012)

INTERVENTIONS:
Other: SEBTC — SEBTC benefits were issued on EBT cards using either the existing EBT delivery systems for the Supplemental Nutrition Assistance Program (SNAP) or Supplemental Nutrition Assistance Program for Women Infants and Children (WIC). Sites selected only one of the two EBT systems to be used to implement SEBTC prior to random assignment; households were not randomized to a specific delivery system.
  Other Names: food assistance; electronic benefit transfer payments
  Arms: $30 SEBTC Benefit Group; $60 SEBTC Benefit Group

SUMMARY:
The Summer Electronic Benefit for Children (SEBTC) demonstration provided food assistance to households with school-aged children during the summer through electronic benefit transfer (EBT) procedures used by the Supplemental Nutrition Assistance Program (SNAP) and Special Supplemental Nutrition Program for Women, Infants and Children (WIC) programs. The evaluation design included two components: an impact study and an implementation study. The evaluation assessed the impact of SEBTC on children's food security and nutritional status, household food expenditures and purchasing behaviors, parental perceptions, and participation in nutrition assistance programs. The implementation study analyzed SEBTC use patterns using administrative data, and described demonstration implementation and costs.

DETAILED DESCRIPTION:
The SEBTC evaluation took place in the summers of 2011 through 2014. Ten grantees implemented the demonstration in a total of 16 sites; the number of participating sites and/or the evaluation components differed by year. In 2011, 5 grantees with five sites participated and the evaluation included implementation and cost analysis, EBT analysis, and an impact study. In 2012, 10 grantees implemented SEBTC in 14 sites and the evaluation included the same study components. In 2013, four grantees with six sites participated and the study components included EBT analysis and an impact study (no implementation or cost data collection). Finally, in 2014, three grantees participated in three sites and only implementation data were collected. Information on human subjects was collected for the evaluation's impact evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Households with children who were certified to receive the National School Lunch program or the School Breakfast Program in the prior school year in participating sites, Summers 2011-2013

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 85000 (Actual)
Dates: Start 2011-01; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Very low food security among children according to the U.S. Household Food Security Survey Module, 30-day reference period | Between 30 and 120 days after SEBTC benefits were issued
  The food intake of any child in the household is reduced and their normal eating patterns are disrupted because the household lacks money and other resources for food

SECONDARY OUTCOMES:
Food insecurity among children according to the U.S. Household Food Security Survey Module, 30-day reference period | Between 30 and 120 days after SEBTC benefits were issued
  Any child in the household experienced very low food security or experienced reduced quality, variety, or desirability of diet.
Children's fruit and vegetable consumption | Between 30 and 120 days after SEBTC benefits were issued
  Average daily cup equivalents of fruit and vegetables
Children's fruit and vegetable consumption without fried potatoes | Between 30 and 120 days after SEBTC benefits were issued
  Average daily cup equivalents of fruit and vegetables, excluding fried potatoes
children's whole grain consumption | between 30 and 120 days after SEBTC benefits were issued
  Average daily consumption of whole grains (in ounces)
Children's dairy consumption | Between 30 and 120 days after SEBTC benefits were issued
  Average daily dairy consumption cup equivalents
Children's consumption of low- and non-fat milk | Between 30 and 120 days after SEBTC benefits were issued
  Any milk consumed was low- or non-fat
Children's consumption of added sugars | Between 30 and 120 days after SEBTC benefits were issued
  Average daily consumption of added sugars (in teaspoons)
Children's consumption of added sugars excluding cereals | Between 30 and 120 days after SEBTC benefits were issued
  Average daily consumption of added sugars excluding cereals (in teaspoons)
Children's consumption of sugar-sweetened beverages | Between 30 and 120 days after SEBTC benefits were issued
  Average daily consumption of sugars (in teaspoons) from sugar-sweetened beverages

OTHER OUTCOMES:
Participation in SNAP | Between 30 and 120 days after SEBTC benefits were issued
  Household participation in the Supplemental Nutrition Assistance Program
Participation in WIC | Between 30 and 120 days after SEBTC benefits were issued
  Household participation in the Special Supplemental Nutrition Assistance Program for Women, Infants and Children
Food expenditures | Between 30 and 120 days after SEBTC benefits were issued
  Total food expenditures from all sources (e.g., cash, SNAP, SEBTC)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bell, Ph.D., Principal Investigator — Abt Associates; Ronette Briefel, Principal Investigator — Mathematica Policy Research, Inc.

IPD SHARING:
Plan to Share IPD: Yes
Contract deliverables include restricted and public use data sets

REFERENCES:
- [Background] Briefel R, Collins A, Bellotti J, Klerman J, Logan CW, Cabili C, Rowe G, Greece J, Owens C, Weiss A. 2011. Congressional Status Report: Summer Electronic Benefits Transfer for Children Demonstrations. Alexandria, V: U.S. Department of Agriculture, Food and Nutrition Service.
- [Background] Briefel R, Collins A, Rowe G, Wolf A, Klerman JA, Logan CW, Wulsin CS, Enver A, Owens C, Jacobson J, Bell S. 2012. Summer Electronic Benefits Transfer for Children (SEBTC) Demonstration: 2012 Congressional Status Report. Alexandria, VA: U.S. Department of Agriculture, Food and Nutrition Service.
- [Result] Collins A, Briefel R, Klerman JA, Rowe G, Wolf A, Logan CW, Gordon A, Wolfson C, Enver A, l Owens C, Cabili C, Bell S. 2013. Summer Electronic Benefits Transfer for Children (SEBTC) Demonstration: Evaluation Findings for the Full Implementation Year. Alexandria, VA: U.S. Department of Agriculture, Food and Nutrition Service
- [Result] Collins AM, Briefel R, Klerman JA, Wolf A, Rowe G, Enver A, Logan CW, Fatima S, Komarovksy M, Lyskawa J, Bell S. 2014. Summer Electronic Benefits Transfer for Children (SEBTC) Demonstration: Findings for the Third Implementation Year. Alexandria, VA: U.S. Department of Agriculture, Food and Nutrition Service.
- [Result] Collins A, Briefel R, Klerman JA, Bell S, Belotti J, Logan C, Gordon A, Wolfe A, McLaughlin S, Enver A, Fernandes M, Wolfson C, Komorovsky M, Cabili C, Owens, C. 2012. Summer EBT for Children Demonstration: Evaluation Findings for the Proof of Concept Year. Alexandria, VA: U.S. Department of Agriculture, Food and Nutrition Service.
- [Result] Collins AM, Briefel, R, Klerman JA, Rowe G, Wolf A, Logan C, Enver A, Fatima S, Gordon A, Lyskawa A. (2016). Summer Electronic Benefits for Children Demonstration: Summary Report. Alexandria, VA: U.S. Department of Agriculture, Food and Nutrition Service.
- [Derived] Collins AM, Klerman JA, Briefel R, Rowe G, Gordon AR, Logan CW, Wolf A, Bell SH. A Summer Nutrition Benefit Pilot Program and Low-income Children's Food Security. Pediatrics. 2018 Apr;141(4):e20171657. doi: 10.1542/peds.2017-1657. PMID 29592869